CLINICAL TRIAL: NCT06508489
Title: A Phase 1/Phase 2, Randomized, Open-label, Multi Cohort, Multi Center, Study Assessing the Safety, Tolerability and Preliminary Efficacy of SAR443579 a Natural Killer Cell Engager (NKCE) Targeting CD123, Administered With Different Agents in Participants With CD123 Expressing Hematological Malignancies
Brief Title: A Study to Investigate Natural Killer Cell Engager (SAR443579) With Different Agents in Participants With Hematological Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Early discontinuation based on strategic sponsor decision not driven by any safety concerns
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD17796; U1111-1280-6173 (Registry Identifier: ICTRP); 2023-509438-20 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-06-27; First posted 2024-07-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Substudy 01: SAR443579 + azacitidine + venetoclax (Experimental): Part 1: Safety run-in: SAR443579 treatment will begin with an identified starting dose. Safety run-in will proceed according to the incidence of DLTs.
  Interventions: Biological: SAR443579; Drug: venetoclax; Drug: azacitidine

INTERVENTIONS:
Biological: SAR443579 — Pharmaceutical form: Powder for solution for infusion Route of administration: intravenous infusion
Drug: venetoclax — Pharmaceutical form :Film coated tablet Route of administration: oral
  Other Names: VENCLYXTO / VENCLEXTA
Drug: azacitidine — Pharmaceutical form: Lyophilized powder for suspension for injection Route of administration: intravenous or subcutaneous

SUMMARY:
This is a parallel, Phase 1/Phase 2, randomized, open label, multi-cohort, multi-center study assessing the safety, tolerability and preliminary efficacy of SAR443579 with different agents for treatment in adolescent and/or adult participants with CD123 expressing hematological malignancies.

This protocol is structured as a master protocol (containing common protocol elements). Individual sub-studies will explore SAR443579 with combination partners, which may include approved or investigational agents.

Experimental sub-studies will be tested through 3 parts:

Part 1: dose finding (such as dose escalation/ safety run-in). Part 2: dose optimization (when applicable). Part 3: dose expansion. In each sub-study, a dose escalation will identify preliminary recommended dose for expansion (pRDE) of SAR443579 and its respective combination partner. Following the determination of the preliminary RDE, additional participants will be enrolled in the dose expansion part, or if dose optimization needs to be further evaluated, additional participants will be enrolled in the "dose optimization/expansion" part. Dose optimization and dose expansion part could involve randomization depending on specific sub-study design.

Study will consist of a screening period, treatment period, and follow-up period.

Participants will receive study treatment until documented disease progression, unacceptable adverse events, participant's decision to stop study treatment, or completion of the maximum cycles allowed in the sub-studies, or the participant meets other criteria for discontinuation per study protocol (whichever occurs first).

DETAILED DESCRIPTION:
Substudy 01:

Title: A Phase 1/Phase 2, open-label, multi-center study, assessing the safety, tolerability and the preliminary efficacy of SAR443579 administered in combination with azacitidine + venetoclax in adult participants with CD123 expressing newly diagnosed Acute Myeloid Leukemia (ND-AML) that are ineligible for intensive chemotherapy

Short title: A study to investigate natural killer cell engager (SAR443579) in combination with azacitidine + venetoclax in adult participants with newly diagnosed acute myeloid leukemia

The expected duration of the study for a participant is approximately about 2.5 years. The study duration includes a screening period, an induction and maintenance. After the end of study treatment participants will enter the follow-up period for up to 2 years.

Planned number of participants:

22 participants planned to be screened, 8 being adults and 14 being elderly; 9-18 participants planned to be enrolled (dose escalation part)

Enrollment will be paused upon completion of Part 1: Dose Escalation. The available data will be reviewed and the recommended doses and schedule for optimization will be selected by the study board. Enrollment in the Part 2: Dose optimization and Part 3: Dose expansion will be provided in a future protocol amendment.

ELIGIBILITY:
Inclusion Criteria:

- Participants with CD123-expressing hematological neoplasm per the 5th edition of the WHO Classification of Hematolymphoid Tumors.

Substudy 01:

* Participants must be ≥18 years of age
* Confirmed diagnosis of Acute Myeloid Leukemia
* Ineligible for intensive chemotherapy. Ineligible for intensive chemotherapy is defined by the following criteria:

A) ≥ 75 years of age, OR

B) 18 to 74 years of age and meeting one or more of the following:

1. Eastern Cooperative Oncology Group (ECOG) performance status 2-3.
2. Cardiac history of congestive heart failure (CHF) requiring treatment or left ventricular ejection fraction (LVEF) ≤50% or symptomatic coronary heart disease confirmed by coronarography or cardiac imaging.
3. Diffusing capacity of the lungs for carbon monoxide (DLCO) ≤65% or forced expiratory volume (FEV1) ≤65%.
4. Creatinine clearance ≥30 to <45 mL/min calculated by modification of diet in renal disease (MDRD) formula.
5. Moderate hepatic impairment with total bilirubin >1.5 to ≤3.0x upper limit of normal (ULN).

   * Subject with an Eastern Cooperative Oncology Group (ECOG) performance status as follows:

a) 0 to 2 for participants ≥75 years of age or b) 0 to 3 for participants 18 to 74 years of age.

* For participants ≥75 years of age, adequate renal function demonstrated by a creatinine clearance ≥30 mL/min, calculated by modification of diet in renal disease (MDRD)
* Subject with adequate liver function demonstrated by the following:

  1. For participants 18 to 74 years of age, aspartate aminotransferase (AST) ≤3.0 × ULN, alanine aminotransferase (ALT) ≤3.0 × ULN and bilirubin ≤3.0 × ULN, unless considered due to leukemic organ involvement ˂5 × ULN.
  2. For participants ≥75 years of age, aspartate aminotransferase (AST) ≤3.0 × ULN, alanine aminotransferase (ALT) ≤3.0 × ULN and bilirubin ≤1.5 × ULN, unless considered due to leukemic organ involvement ˂5 × ULN.

Exclusion Criteria:

* Any clinically significant, uncontrolled medical conditions (including any serious active systemic infection that is not controlled)
* Known second malignancy either progressing or requiring active treatment within the last 3 years prior to first IMP administration
* Known acquired immunodeficiency syndrome (AIDS-related illnesses) or HIV disease requiring antiretroviral treatment, or having active hepatitis B or C infection, or SARS-CoV-2 infection. With exception for:

  1. HBV as determined by positive test for hepatitis B surface antigen (HBsAg) and/or HBV DNA. Participant who tests positive for anti-hepatitis B core (HBc) antigen IgG (with or without testing positive for anti-HBs), but tests negative for HBsAg and HBV DNA, is eligible.
  2. A participant who tests positive for anti-HCV antibodies and has undetectable HCV RNA without receiving antiviral treatment for HCV is eligible.
* Active, known, or suspected clinically significant autoimmune disease that has required systemic treatment in the past 2 years prior to first IMP administration, except controlled by replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc)
* Predicted life expectancy ≤3 months.
* Medical conditions requiring treatment with medications with narrow therapeutic index that are substrates of CYP enzymes and that cannot be closely monitored to allow for dose adjustment.
* Ongoing adverse event of NCI CTCAE [Version 5.0] Grade 2 or greater severity cause by any prior anti-cancer therapy

Substudy 01:

* Patient with Acute Promyelocytic Leukemia (APL)
* Known active central nervous system involvement with AML at the time of enrollment as evidenced by cytology or pathology
* Cardiovascular disease of New York Heart Association (NYHA) Class ≥2.
* Malabsorption syndrome or other condition that precludes enteral route of administration
* A baseline QTc interval of (using the Fridericia correction calculation) >470 msec.
* Subject has received treatment with at least one of the following:

  1. A hypomethylating agent, venetoclax and/or chemo therapeutic agent for AML other than hydroxyurea used for disease control prior to the initiation of study therapy.
  2. Experimental therapies for AML.
  3. Concomitant medications of strong and moderate CYP3A inducers within 7 days prior to the initiation of study treatment.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs)/serious adverse events (SAEs)/adverse events of special interest (AESIs), laboratory abnormalities | Day 1 to 30 days after the last administration of study treatment
Substudy 01: Incidence of dose limiting toxicities (DLTs) (escalation part) | Day 1 to Day 28
Substudy 01: Complete Remission (CR) rate (optimization part) | Day 1 to 30 days after the last administration of study treatment
  Proportion of participants who have a CR (Complete Remission) determined by the Investigator according to 2022 European Leukemia Net (ELN) recommendations for diagnosis and management of AML
Substudy 01: Complete Remission (CR) rate (expansion part) | Day 1 up to 6 months
  Proportion of participants who have a CR (Complete Remission) determined by the Investigator according to 2022 European Leukemia Net (ELN) recommendations for diagnosis and management of AML

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs) and clinically significant laboratory abnormalities (expansion part) | Day 1 to 30 days after the last administration of study treatment
  According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) V 5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading for cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS)
Incidence of anti-drug anti body (ADA) against SAR443579 | Day 1 to 30 days after the last administration of study treatment
Substudy 01: Percentage of participants with Minimal residual disease (expansion part) | Day 1 up to 6 months
  As defined by 2022 ELN recommendations for AML
Substudy 01: Pharmacokinetic (PK) parameter of SAR443579: Ctrough | Day 1 up to 10 cycles (each cycle 28 days)
  Concentrations observed at the end the dosing period during repeated administration for SAR443579
Substudy 01: PK parameter of venetoclax: Cmax | Day 1 to Day 28
  Maximum concentration observed for venetoclax
Substudy 01: PK parameter of azacitidine: Cmax | Day 1 to Day 28
  Maximum concentration observed for azacitidine
Substudy 01: PK parameter of venetoclax: AUC | Day 1 to Day 28
  Area under the blood concentration versus time curve extrapolated to infinity for venetoclax
Substudy 01: PK parameter of azacitidine: AUC | Day 1 to Day 28
  Area under the blood concentration versus time curve extrapolated to infinity for azacitidine
Substudy 01: Composite Complete Remission (CRc) rate | Day 1 up to 6 months
  Proportion of participants who have a CR (Complete Remission) + CRh (complete remission with partial hematologic recovery) + CRi (Complete Remission with Incomplete Hematologic Recovery) determined by the Investigator according to 2022 European Leukemia Net (ELN) recommendations for diagnosis and management of AML.
  (CRc = CR + CRh + CRi)
Substudy 01: Overall response rate (expansion part) | Day 1 up to 6 months
  Proportion of participants who have a CR or CRi or CRh or PR or MLFS (morphological leukemia-free state) according to the 2022 ELN criteria.
Substudy 01: Duration of CR (expansion part) | Day 1 up to 24 months after the last administration from study treatment
  Defined as the time interval from the first documented evidence of CR until disease relapse as per 2022 ELN recommendations or death due to any cause, whichever comes first
Substudy 01: Duration of CRc (expansion part) | Day 1 up to 24 months after the last administration from study treatment
  Defined as the time interval from first documented evidence of CRc (CR, CRh or CRi) until disease relapse as per 2022 ELN recommendations or death due to any cause, whichever comes first
Substudy 01: Duration of overall response (expansion part) | Day 1 up to 24 months after the last administration from study treatment
  Defined as the time from the first documented evidence of CR or CRi or CRh or PR or MLFS until disease relapse as per 2022 ELN recommendations or death due to any cause, whichever comes first
Substudy 01: Alternative CR rate (expansion part) | Day 1 up to 6 months
  Defined as the proportion of participants with CR+CRh (complete remission with partial hematological recovery)
Substudy 01: Duration of alternative CR (expansion part) | Day 1 up to 24 months after the last administration from study treatment
  Defined as the time from the first documented evidence of CR or CRh until disease relapse as per 2022 ELN recommendations or death due to any cause, whichever comes first
Substudy 01: Event-free survival (EFS) (expansion part) | Day 1 up to 24 months after the last administration from study treatment
  Defined as the time interval from the first day of treatment assignment to the date of earliest evidence of relapse, treatment failure, or death
Substudy 01: Overall survival (expansion part) | Day 1 up to 24 months after the last administration from study treatment
  Defined as time interval from the first day of treatment assignment to death from any cause
Substudy 01: Rate of hematopoietic stem cell transplantation (HSCT) procedures immediately following study treatment administration but prior to subsequent therapy for treatment of AML (all parts) | Day 1 up to 24 months after the last administration from study treatment
  The HSCT rate is defined as the proportion of such participants who undergo HSCT through study treatment but before subsequent therapy, among the safety/exposed population
Substudy 01: Time to treatment failure (TTF) (expansion part) | Day 1 up to 24 months after the last administration from study treatment
  Defined as the time from first day of treatment assignment to discontinuation for any reason excluding remission, for example relapsed disease, refractory disease, unacceptable AE, participant preference or death
Substudy 01: Rate of conversion from transfusion dependence to transfusion independence (all parts) | Day 1 to Day 56
  The transfusion dependency (TD) at baseline is based on the receipt of any red blood cell or platelets transfusions within at least 28 days prior to the start of study treatment. For post baseline treatment, transfusion independency (TI) will be defined as the absence of transfusion during any 56 consecutive day period during treatment.
Substudy 01: Rate of participants who are transfusion independent at baseline and remain independent during 56-day post-baseline period (all parts) | Day 1 to Day 56
  Transfusion independency (TI) will be defined as the absence of transfusion during any 56 consecutive day period during treatment.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - City of Hope National Medical Center- Site Number : 8400003, Duarte, California
  - Montefiore Medical Center - Moses Campus- Site Number : 8400004, The Bronx, New York
  - The Ohio State University Wexner Medical Center - Ohio State Outpatient Care Upper Arlington- Site Number : 8400001, Columbus, Ohio
  - Oregon Health and Science University- Site Number : 8400006, Portland, Oregon
  - The University of Texas MD Anderson Cancer Center- Site Number : 8400008, Houston, Texas
- Australia (2):
  - Investigational Site Number : 0360002, Wollongong, New South Wales
  - Investigational Site Number : 0360001, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org